CLINICAL TRIAL: NCT00001074
Title: A Phase I/II Dosing Study of the Safety and Antiretroviral Activity of Hydroxyurea Alone and in Combination With ddI Compared With ddI Alone in Subjects With HIV Infection
Brief Title: The Safety and Effectiveness of Hydroxyurea and ddI Used Individually or Together in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 307; 11282 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Antiviral Agents; Hydroxyurea
MeSH Terms: conditions — HIV Infections | interventions — Hydroxyurea; Didanosine

INTERVENTIONS:
Drug: Hydroxyurea
Drug: Didanosine

SUMMARY:
To determine the safety and tolerability of hydroxyurea at two doses alone and in combination with didanosine (ddI). To compare the short term antiviral effect of ddI monotherapy versus hydroxyurea plus ddI, as measured by plasma RNA levels at 8 weeks of therapy. [AS PER AMENDMENT 10/1/97: Accrual to arms involving hydroxyurea alone has been closed.] Current antiviral therapies for HIV-1 are limited by a few choices, and the lack of sustained clinical benefit from the drugs. The mechanisms that account for the lack of prolonged inhibition of viral replication by these agents are not fully understood. The activity of RT inhibitors might be potentiated by inhibiting host cellular enzymes essential for efficient HIV reverse transcription. Based on this information, comparisons of the antiviral effects of ddI monotherapy and hydroxyurea plus ddI, with the cellular enzyme ribonucleotide reductase as a potential target, should be done.

DETAILED DESCRIPTION:
Current antiviral therapies for HIV-1 are limited by a few choices, and the lack of sustained clinical benefit from the drugs. The mechanisms that account for the lack of prolonged inhibition of viral replication by these agents are not fully understood. The activity of RT inhibitors might be potentiated by inhibiting host cellular enzymes essential for efficient HIV reverse transcription. Based on this information, comparisons of the antiviral effects of ddI monotherapy and hydroxyurea plus ddI, with the cellular enzyme ribonucleotide reductase as a potential target, should be done.

This is a 24-week study, with two 12-week treatment periods. Patients are randomized to one of five treatment arms based upon a patient's history of antiretroviral therapy (naive vs. experienced). The five treatment arms are:

1. ddI plus hydroxyurea placebo.
2. hydroxyurea (lower dose) plus ddI placebo for 4 weeks; then hydroxyurea (higher dose) plus ddI.
3. hydroxyurea (higher dose) plus ddI placebo for 4 weeks; then hydroxyurea (higher dose) plus ddI.
4. hydroxyurea (lower dose) plus ddI.
5. hydroxyurea (higher dose) plus ddI. After the completion of week 12, patients on combination therapy remain on their current therapy and patients on ddI plus placebo have hydroxyurea replace the placebo at 1 of 2 assigned doses (1:1 randomization). AS PER AMENDMENT 5/5/97: If after the 24-week treatment period, a patient has an RNA level less than or equal to 5,000 copies/ml or less than 20,000 copies/ml with a greater than 1 log10 decline from baseline, she has the option to continue therapy open-label ddI plus hydroxyurea for an additional 24 weeks.

AS PER AMENDMENT 10/1/97: Accrual to the arms involving hydroxyurea alone has been closed. Patients are randomized to one of the three treatment arms, as follows:

1. hydroxyurea placebo plus ddI.
2. hydroxyurea (lower dose) plus ddI.
3. hydroxyurea (higher dose) plus ddI.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

AS PER AMENDMENT 5/5/97:

* PCP prophylaxis with trimethoprim/sulfamethoxazole or Dapsone.

Patients must have:

* HIV-1 infection.
* AS PER AMENDMENT 5/5/97:
* CD4 count of 200 - 700 cells/mm3 within 60 days prior to study entry.
* AS PER AMENDMENT 10/1/97:
* HIV RNA plasma level < 20,000 copies/ml within 60 days of enrollment (obtained at a laboratory certified to perform the Roche Monitor assay).

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* CMV, MAC, toxoplasmosis, or disseminated fungal infection requiring acute or chronic therapy.
* Significant medical illness as determined by investigator.
* Active diagnosis of any malignancy, including visceral Kaposi's sarcoma or extensive cutaneous Kaposi's sarcoma for which systemic chemotherapy is anticipated within the next 24 weeks.
* Current Grade 2 or greater peripheral neuropathy.

Concurrent Medication:

Excluded:

* Acute or chronic therapy for CMV, MAC, toxoplasmosis, or disseminated fungal infection.

AS PER AMENDMENT 5/5/97:

* All antiretroviral medications other than those provided on study.
* Systemic chemotherapy for active malignancies, including systemic treatment for KS.
* Agents with myelosuppressive potential, including tegretol, carboplatin, carmustine, cyclophosphamide and fluorouracil.
* Granulocyte colony stimulating factor (G-CSF) except while hydroxyurea or matching placebo is held.

Drugs associated with peripheral neuropathy, including:

* hydralazine, disulfiram, nitrofurantoin, cisplatinum, diethyldithiocarbamate, gold, rifampin, chloramphenicol, clioquinol, ethambutol, ethionamide, glutethimide, sodium cyanate, and thalidomide.

Patients with any of the prior conditions are excluded:

* History of transfusion dependent anemia, defined as any history of repeated transfusion with two or more units of red blood cells.
* At the discretion of the investigator, history of pancreatitis.

Prior Medication:

Excluded:

* More than 2 weeks prior treatment with ddI.

AS PER AMENDMENT 5/5/97:

* Other antiretrovirals must be discontinued at least 14 days prior to randomization.
* Prior hydroxyurea.
* Any candidate HIV vaccine or agent with potential immune modulating effects within the past 30 days.
* Any colony stimulating factor or erythropoietin within the past 60 days.

Prior Treatment:

Excluded:

* Transfusion with red blood cells within the past 60 days.

Risk Behavior:

Excluded:

* At the investigator's discretion, any active substance abuse, including alcohol abuse interfering with compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Study Completion 2000-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Frank, MD, Study Chair — Division of Infectious Diseases, University of Pennsylvania; Joseph Eron, MD, Study Chair — University of North Carolina
Locations (18):
- United States (18):
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Stanford Univ Med Ctr, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Result] Frank I, Boucher H, Fiscus S, Flexner C, Valentine F, Gulick R, Fox L, Eron J. Phase I/II dosing study of once-daily hydroxyurea (HU) alone vs didanosine (ddI) alone vs ddI + HU. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:143 (abstract no 402)
- [Result] Frank I, Bosch RJ, Fiscus S, Valentine F, Flexner C, Segal Y, Ruan P, Gulick R, Wood K, Estep S, Fox L, Nevin T, Stevens M, Eron JJ Jr; ACTG 307 Protocol Team. Activity, safety, and immunological effects of hydroxyurea added to didanosine in antiretroviral-naive and experienced HIV type 1-infected subjects: a randomized, placebo-controlled trial, ACTG 307. AIDS Res Hum Retroviruses. 2004 Sep;20(9):916-26. doi: 10.1089/aid.2004.20.916. PMID 15597521